CLINICAL TRIAL: NCT04264403
Title: Effect of Renal Denervation on Blood Pressure in Patients With Chronic Kidney Disease and Uncontrolled Hypertension
Brief Title: Renal Denervation in Chronic Kidney Disease - RDN-CKD Study
Acronym: RDN-CKD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Erlangen-Nürnberg Medical School (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: RDN2019CKD
Record Dates: First submitted 2020-01-31; First posted 2020-02-11 (Actual); Last update posted 2023-12-21 (Actual); Status verified 2023-11

CONDITIONS: Uncontrolled Hypertension; Renal Denervation; Chronic Kidney Disease stage3
Keywords: Chronic Kidney Disease; Renal Denervation; Uncontrolled Hypertension
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Intervention Model Description: RDN-CKD Study is a prospective, randomized (1:1, central randomization), double-blind (unblinded interventionalist and blinded study team at each center), sham controlled, multicenter feasibility study.
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: The subjects and all study personnel taking BP measurements will be blinded to the randomization. Subjects will complete a blinding assessment prior to hospital pre-discharge and at 3 weeks, 6 months and 12 months FU.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Renal Denervation (Active Comparator): All subjects will undergo a diagnostic, renal angiogram (based on clinical grounds to rule out renal artery stenosis) which should be per Institutional practice via femoral artery access. Randomization will occur following the diagnostic renal angiogram. If randomized to the Renal Denervation Group RDN procedure will be applied using the Paradise® Renal Denervation System. The Paradise® Renal Denervation System is a catheter-based device designed to use ultrasound energy to thermally ablate the afferent and efferent nerves surrounding the renal artery and serving the kidney.
  Interventions: Device: Renal denervation
- Sham Procedere (No Intervention): All subjects will undergo a diagnostic, renal angiogram (based on clinical grounds to rule out renal artery stenosis) which should be per Institutional practice via femoral artery access. Randomization will occur following the diagnostic renal angiogram. In these patients no RDN will be performed.

INTERVENTIONS:
Device: Renal denervation — The Paradise® Renal Denervation System (Paradise System) is CE-marked in countries accepting the CE mark. The system is a catheter-based device designed to use ultrasound energy to thermally ablate the afferent and efferent nerves surrounding the renal artery and serving the kidney.
  Arms: Renal Denervation

SUMMARY:
RDN-CKD Study is a prospective, randomized (1:1, central randomization), double-blind (unblinded interventionalist and blinded study team at each center), sham controlled, multicenter feasibility study. The purpose of the RDN-CKD Study is to demonstrate that renal denervation (RDN) effectively reduces 24-h ambulatory BP in 80 patients with chronic kidney disease (CKD) stage 3a or 3b.

DETAILED DESCRIPTION:
1. Introduction Uncontrolled hypertension is more prevalent in patients with chronic kidney disease (CKD) and the risk of developing end-stage renal disease is increased in patients with uncontrolled hypertension. Clinical and experimental studies have clearly shown that sympathetic nerve activity is increased in CKD and substantially aggravates the progression of CKD. Recent clinical studies have indicated that invasive, catheter-based renal denervation (RDN) decreases the sympathetic nerve activity in the whole body and in particular in the kidneys. In patients with primary hypertension washed off of antihypertensive medications, RDN has been found to significantly decrease blood pressure (BP) in two randomized, double blind, sham-controlled studies.
2. Study Purpose The purpose of the RDN-CKD Study is to demonstrate that RDN effectively reduces 24-h ambulatory BP in patients with CKD stage 3.
3. Study Design RDN-CKD Study is a prospective, randomized (1:1, central randomization), double-blind (unblinded interventionalist and blinded study team at each center), sham controlled, multicenter feasibility study. All centers have participated at least in one of the sham-controlled trials in primary hypertension thereby having established an unblinded and a blinded team.
4. Patient Population

80 patients with CKD stages 3a or 3b (according to the currently used estimation formulas [MDRD, CKD-EPI] and uncontrolled hypertension.

5 Endpoints Primary Efficacy Endpoint The primary efficacy endpoint will be the change in systolic 24-h ambulatory BP at 6 months post-procedure compared between the 2 groups.

6 Visit and Follow-Up Schedule The primary efficacy endpoint will be assessed at 26 weeks (6 months) post-procedure in both cohorts; however, all subjects will be followed for a minimum of 12 months post-procedure. Scheduled in-clinic follow-up (FU) visits will occur at 3, 6, 12 (3 months), 19, 26 (6 months), 39 and 52 (12 months) weeks post procedure.

7 Blinding The subjects and all study personnel taking BP measurements will be blinded to the randomization. Subjects will complete a blinding assessment prior to hospital pre-discharge and at 3 weeks and 6 months FU.

8 Crossover to treatment Crossover of patients allocated to the sham group is allowed after 12 months. At that time, after 12 months of blinded FU, unblinding of the individual patient takes place. To be eligible for crossover treatment, patients have to fulfill the same BP criteria as specified at the inclusion criteria and exclusion criteria within the next 4 weeks after FU.

All randomized patients will be included in a registry after 12 months to capture long-term safety signals.

9 Medication Adherence Adherence to drug therapy will be captured by interviewing patients, checking the patient's BP diary and by urinary toxicological analysis at baseline, 6 months, and 12 months visit.

10 Safety Signals A major combined safety endpoint is the incidence of any major adverse events (MAE) through the 12 months FU.

11 Study Geographies The RDN-CKD Study will be conducted at 4 clinical investigational sites, which are the University Hospitals in Erlangen, Homburg/Saar, Düsseldorf, and Nürnberg.

12 Escape Criteria Enrolled subjects will be excluded if office (attended) BP exceeds ≥170/105 mmHg confirmed by 7-day average of home blood pressure measurements ≥ BP >160/100 mmHg or confirmed by office (attended) BP ≥170/105 mmHg at another study visit.

13 Ethics The study will be conducted in accordance with the declaration of Helsinki, ISO 14155:2011, FDA 21 CFR parts 50, 54, 56, 812 and other applicable local and national regulations.

ELIGIBILITY:
Inclusion Criteria:

* CKD stage 3 (eGFR 30-59 ml/min/1.73m² [according to the currently used estimation formulas: MDRD, CKD-EPI]) with diabetic or non-diabetic nephropathy
* Uncontrolled hypertension with 1-5 drug classes (renin angiotensin system [RAS] blockade is mandatory, unless intolerance to RAS blockers has been documented) and systolic office (attended) BP ≥140 mmHg confirmed by 24-h ambulatory BP systolic ≥130 mmHg
* Patient is adhering to a stable drug regimen including RAS blockade without changes for a minimum of 4 weeks.
* Individual is ≥ 18 years of age, both genders are included.

Exclusion Criteria:

* Anatomically significant renal artery abnormality in either renal artery which in the eyes of the interventionalist would interfere with safe catheter Placement
* Other cause of Hypertension that can be treated by Intervention/surgery (e.g. hemodynamically relevant renal artery stenosis, functional adrenal adenoma)
* Prior renal denervation procedure
* Office (attended) BP ≥ 180 mmHg systolic and/or ≥ 110 mmHg diastolic
* 24-h ambulatory BP ≥ 160 mmHg systolic
* Anatomic or functional solitary kidney, kidney transplantation
* Lack of capturing serum creatinine levels in the past
* Secondary hypertension other than obstructive sleep apnea
* Type 1 diabetes mellitus
* Nephrotic syndrome
* Contraindication to magnetic resonance imaging (MRI)
* Individual has experienced a myocardial infarction, unstable angina pectoris, or a cerebrovascular accident within 3 months of the screening visit
* Acute episode of renal disease requiring uptitration of any immunosuppressive drug regimen within the last 3 months
* Subject is pregnant, nursing, or intends to become pregnant
* Enrollment in another interventional research protocol.
* Any condition that, at the discretion of the investigator, would preclude participation in the study (e.g. non-adherence)

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2020-01-23 (Actual); Primary Completion 2023-12-23 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
change in systolic 24-h ambulatory BP | at 6 month post-procedure
  compared between the 2 groups (updated; please see details in the SAP uploaded)

SECONDARY OUTCOMES:
Change in systolic 24-h ambulatory BP | at 3 and 12 month post-procedure
  compared between the 2 groups (updated; please see details in the SAP uploaded)
Change in diastolic 24-h ambulatory BP at 3, 6 and 12 months post-procedure | at 3, 6 and 12 months post-procedure
  compared between the 2 groups (updated; please see details in the SAP uploaded)
Change in office (attended) systolic and diastolic BP | at 3, 6 and 12 months post-procedure
  between the 2 groups (updated; please see details in the SAP uploaded)
Responder rate in BP (systolic office (attended) BP ≥10 mmHg, 24-h systolic ambulatory BP ≥ 5 mmHg) | at 3, 6 and 12 months post-procedure
  compared between the 2 groups (updated; please see details in the SAP uploaded)
Change in estimated glomerular filtration rate [eGFR] | at 3, 6 and 12 months post-procedure
  compared between the 2 groups (updated; please see details in the SAP uploaded)
Change of the slope of eGFR | after half year and one year post-procedure
  compared between the 2 groups (updated; please see details in the SAP uploaded)
Change of the slope of eGFR | at 1 year post-procedure
  compared to the historical slope the year before (updated; please see details in the SAP uploaded)
Change in albuminuria quantitatively and by category | at 6 and 12 months post-procedure
  compared between the 2 groups (updated; please see details in the SAP uploaded)

CONTACTS AND LOCATIONS:
Overall Officials: Roland E Schmieder, MD, Principal Investigator — Clinical Research Center, Department of Nephrology and Hypertension, University of Erlangen-Nuremberg
Locations (4):
- Germany (4):
  - Heinrich Heine University Düsseldorf, Nephrologie, Germany, Düsseldorf
  - Clinical Research Center, Department of Nephrology and Hypertension, University of Erlangen-Nuremberg, Erlangen
  - Klinik für Innere Medizin III, Kardiologie, Angiologie Und Internistische Intensivmedizin, Saarland University Hospital, Saarland University, Homburg
  - Clinical Research Center Nuremberg, Department of Nephrology, University Hospital Erlangen, Nuremberg

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Klag MJ, Whelton PK, Randall BL, Neaton JD, Brancati FL, Ford CE, Shulman NB, Stamler J. Blood pressure and end-stage renal disease in men. N Engl J Med. 1996 Jan 4;334(1):13-8. doi: 10.1056/NEJM199601043340103. PMID 7494564
- [Background] Chowdhury EK, Langham RG, Ademi Z, Owen A, Krum H, Wing LM, Nelson MR, Reid CM; Second Australian National Blood Pressure Study Management Committee. Rate of change in renal function and mortality in elderly treated hypertensive patients. Clin J Am Soc Nephrol. 2015 Jul 7;10(7):1154-61. doi: 10.2215/CJN.07370714. Epub 2015 Apr 21. PMID 25901093
- [Background] Hering D, Mahfoud F, Walton AS, Krum H, Lambert GW, Lambert EA, Sobotka PA, Bohm M, Cremers B, Esler MD, Schlaich MP. Renal denervation in moderate to severe CKD. J Am Soc Nephrol. 2012 Jul;23(7):1250-7. doi: 10.1681/ASN.2011111062. Epub 2012 May 17. PMID 22595301
- [Background] Veelken R, Schmieder RE. Renal denervation--implications for chronic kidney disease. Nat Rev Nephrol. 2014 Jun;10(6):305-13. doi: 10.1038/nrneph.2014.59. Epub 2014 Apr 15. PMID 24733118
- [Background] Converse RL Jr, Jacobsen TN, Toto RD, Jost CM, Cosentino F, Fouad-Tarazi F, Victor RG. Sympathetic overactivity in patients with chronic renal failure. N Engl J Med. 1992 Dec 31;327(27):1912-8. doi: 10.1056/NEJM199212313272704. PMID 1454086
- [Background] Vonend O, Marsalek P, Russ H, Wulkow R, Oberhauser V, Rump LC. Moxonidine treatment of hypertensive patients with advanced renal failure. J Hypertens. 2003 Sep;21(9):1709-17. doi: 10.1097/00004872-200309000-00021. PMID 12923404
- [Background] Schlaich MP, Bart B, Hering D, Walton A, Marusic P, Mahfoud F, Bohm M, Lambert EA, Krum H, Sobotka PA, Schmieder RE, Ika-Sari C, Eikelis N, Straznicky N, Lambert GW, Esler MD. Feasibility of catheter-based renal nerve ablation and effects on sympathetic nerve activity and blood pressure in patients with end-stage renal disease. Int J Cardiol. 2013 Oct 3;168(3):2214-20. doi: 10.1016/j.ijcard.2013.01.218. Epub 2013 Feb 28. PMID 23453868
- [Background] Ott C, Mahfoud F, Schmid A, Toennes SW, Ewen S, Ditting T, Veelken R, Ukena C, Uder M, Bohm M, Schmieder RE. Renal denervation preserves renal function in patients with chronic kidney disease and resistant hypertension. J Hypertens. 2015 Jun;33(6):1261-6. doi: 10.1097/HJH.0000000000000556. PMID 25923731
- [Background] Oparil S, Schmieder RE. New approaches in the treatment of hypertension. Circ Res. 2015 Mar 13;116(6):1074-95. doi: 10.1161/CIRCRESAHA.116.303603. PMID 25767291
- [Background] Azizi M, Sapoval M, Gosse P, Monge M, Bobrie G, Delsart P, Midulla M, Mounier-Vehier C, Courand PY, Lantelme P, Denolle T, Dourmap-Collas C, Trillaud H, Pereira H, Plouin PF, Chatellier G; Renal Denervation for Hypertension (DENERHTN) investigators. Optimum and stepped care standardised antihypertensive treatment with or without renal denervation for resistant hypertension (DENERHTN): a multicentre, open-label, randomised controlled trial. Lancet. 2015 May 16;385(9981):1957-65. doi: 10.1016/S0140-6736(14)61942-5. Epub 2015 Jan 26. PMID 25631070
- [Background] Townsend RR, Mahfoud F, Kandzari DE, Kario K, Pocock S, Weber MA, Ewen S, Tsioufis K, Tousoulis D, Sharp ASP, Watkinson AF, Schmieder RE, Schmid A, Choi JW, East C, Walton A, Hopper I, Cohen DL, Wilensky R, Lee DP, Ma A, Devireddy CM, Lea JP, Lurz PC, Fengler K, Davies J, Chapman N, Cohen SA, DeBruin V, Fahy M, Jones DE, Rothman M, Bohm M; SPYRAL HTN-OFF MED trial investigators*. Catheter-based renal denervation in patients with uncontrolled hypertension in the absence of antihypertensive medications (SPYRAL HTN-OFF MED): a randomised, sham-controlled, proof-of-concept trial. Lancet. 2017 Nov 11;390(10108):2160-2170. doi: 10.1016/S0140-6736(17)32281-X. Epub 2017 Aug 28. PMID 28859944
- [Background] Mahfoud F, Cremers B, Janker J, Link B, Vonend O, Ukena C, Linz D, Schmieder R, Rump LC, Kindermann I, Sobotka PA, Krum H, Scheller B, Schlaich M, Laufs U, Bohm M. Renal hemodynamics and renal function after catheter-based renal sympathetic denervation in patients with resistant hypertension. Hypertension. 2012 Aug;60(2):419-24. doi: 10.1161/HYPERTENSIONAHA.112.193870. Epub 2012 Jun 25. PMID 22733462
- [Background] Mahfoud F, Schmieder RE, Azizi M, Pathak A, Sievert H, Tsioufis C, Zeller T, Bertog S, Blankestijn PJ, Bohm M, Burnier M, Chatellier G, Durand Zaleski I, Ewen S, Grassi G, Joner M, Kjeldsen SE, Lobo MD, Lotan C, Luscher TF, Parati G, Rossignol P, Ruilope L, Sharif F, van Leeuwen E, Volpe M, Windecker S, Witkowski A, Wijns W. Proceedings from the 2nd European Clinical Consensus Conference for device-based therapies for hypertension: state of the art and considerations for the future. Eur Heart J. 2017 Nov 21;38(44):3272-3281. doi: 10.1093/eurheartj/ehx215. No abstract available. PMID 28475773
- [Background] Krum H, Schlaich MP, Sobotka PA, Bohm M, Mahfoud F, Rocha-Singh K, Katholi R, Esler MD. Percutaneous renal denervation in patients with treatment-resistant hypertension: final 3-year report of the Symplicity HTN-1 study. Lancet. 2014 Feb 15;383(9917):622-9. doi: 10.1016/S0140-6736(13)62192-3. Epub 2013 Nov 7. PMID 24210779
- [Background] Kandzari DE, Bohm M, Mahfoud F, Townsend RR, Weber MA, Pocock S, Tsioufis K, Tousoulis D, Choi JW, East C, Brar S, Cohen SA, Fahy M, Pilcher G, Kario K; SPYRAL HTN-ON MED Trial Investigators. Effect of renal denervation on blood pressure in the presence of antihypertensive drugs: 6-month efficacy and safety results from the SPYRAL HTN-ON MED proof-of-concept randomised trial. Lancet. 2018 Jun 9;391(10137):2346-2355. doi: 10.1016/S0140-6736(18)30951-6. Epub 2018 May 23. PMID 29803589
- [Background] Azizi M, Schmieder RE, Mahfoud F, Weber MA, Daemen J, Davies J, Basile J, Kirtane AJ, Wang Y, Lobo MD, Saxena M, Feyz L, Rader F, Lurz P, Sayer J, Sapoval M, Levy T, Sanghvi K, Abraham J, Sharp ASP, Fisher NDL, Bloch MJ, Reeve-Stoffer H, Coleman L, Mullin C, Mauri L; RADIANCE-HTN Investigators. Endovascular ultrasound renal denervation to treat hypertension (RADIANCE-HTN SOLO): a multicentre, international, single-blind, randomised, sham-controlled trial. Lancet. 2018 Jun 9;391(10137):2335-2345. doi: 10.1016/S0140-6736(18)31082-1. Epub 2018 May 23. PMID 29803590
- [Background] Ott C, Schmid A, Ditting T, Veelken R, Uder M, Schmieder RE. Effects of renal denervation on blood pressure in hypertensive patients with end-stage renal disease: a single centre experience. Clin Exp Nephrol. 2019 Jun;23(6):749-755. doi: 10.1007/s10157-019-01697-7. Epub 2019 Feb 19. PMID 30783914
- [Derived] Abid S, Mehta S, Munazzah F, Yager N, Baloch S, Hongalgi K. Renal Denervation: A New Era in the Management of Resistant Hypertension. Kidney360. 2025 Nov 1;6(11):2010-2016. doi: 10.34067/KID.0000000961. Epub 2025 Aug 13. PMID 40802676

DOCUMENTS (1):
  • Statistical Analysis Plan (2023-09-01): https://cdn.clinicaltrials.gov/large-docs/03/NCT04264403/SAP_000.pdf